CLINICAL TRIAL: NCT00498745
Title: A Single Dose Bioavailability Study of 2 New Formulations of HKI-272 (240 mg) Compared With a Reference Capsule and an Oral Solution in Healthy Adult Subjects
Brief Title: Study Comparing 2 New Formulations of HKI-272 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 3144A1-1109
Record Dates: First submitted 2007-07-09; First posted 2007-07-10 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
MeSH Terms: interventions — neratinib

INTERVENTIONS:
Drug: neratinib — HKI-272

SUMMARY:
To evaluate the comparative bioavailability of 2 new tablet formulations of HKI-272 with a reference capsule and an oral solution in healthy subjects.

ELIGIBILITY:
Criteria:

* Healthy male and female subjects aged 18 to 50 years.
* Women of nonchildbearing potential (WONCBP)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36
Dates: Start 2007-07; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The data from this study along with in vitro data will be used to explore in vitro/in vivo correlation for HKI-272 to support formulation development.

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (1):
- San Antonio, Texas, United States